CLINICAL TRIAL: NCT05889494
Title: Autologous Whole Blood Management for Reduction of Blood Product Transfusion in Adult Cardiac Surgery Patients: a Local Feasibility/Pilot Study
Brief Title: Autologous Whole Blood Management for Transfusion Reduction in Adult Cardiac Surgery Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: University Hospital Foundation (Other); Alberta Innovates Health Solutions (Other); EPICORE Centre (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00110883
Record Dates: First submitted 2023-05-04; First posted 2023-06-05 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Postoperative Hemorrhage; Postoperative Anemia; Postoperative Blood Loss
Keywords: Cardiac surgery; Postoperative coagulopathy; Autologous whole blood transfusion; Acute normovolemic hemodilution; Intraoperative autologous transfusion
MeSH Terms: conditions — Postoperative Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The participant, intensive care unit physician, and outcome assessors will be blinded to study arm. The intraoperative anesthesiologist will not be blinded to study arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous Whole Blood Management (Experimental): Intraoperative high volume autologous whole blood withdrawal prior to cardiopulmonary bypass (CPB) with re-transfusion following weaning from CPB.
  Interventions: Other: Autologous Whole Blood Management
- Allogenic and Derivative Transfusion (Active Comparator): Control arm participants will receive standard care involving transfusion of plasma, platelets, cryoprecipitate, and/or lyophilized concentrates following weaning from CPB.
  Interventions: Other: Standard Care involving allogenic and/or derivative transfusion.

INTERVENTIONS:
Other: Autologous Whole Blood Management — Intraoperative high volume autologous whole blood withdrawal with re-transfusion following weaning from CPB.
  Other Names: Intraoperative autologous whole blood donation
  Arms: Autologous Whole Blood Management
Other: Standard Care involving allogenic and/or derivative transfusion. — Therapeutic treatment of CPB-induced coagulopathy using donated allogenic blood products including plasma, platelets, and cryoprecipitate and/or derivative administration using prothrombin complex and fibrinogen concentrates.
  Arms: Allogenic and Derivative Transfusion

SUMMARY:
The goal of this pilot trial is to test a protocol for a planned Canada-wide clinical trial looking at whether or not the use of a patients own blood works as good as the current standard of care using donated blood products to reduce blood loss in adult patients having heart surgery.

The main questions this study aims to answer are:

* Is the protocol practical, effective, and efficient.
* Does the use of a patients own blood lower the following: bleeding, the amount donated blood products given, and complications.

Participants will be separated into two groups by a process that is like flipping a coin. One group will donate blood to themselves in the operating room and get their own blood back after surgery. The other group will be given blood products donated by other humans to treat the bleeding after heart surgery.

Researchers will compare both groups to see if patients that get their own blood have fewer donated blood products given at time of heart surgery and have less complications after surgery.

DETAILED DESCRIPTION:
Cardiac surgery patients are at risk for perioperative bleeding and transfusion due to the invasiveness of the surgery and an acquired coagulopathy that is unique to this sub-specialty. High transfusion rates in this population are related to surgical field blood loss and the development of a multi-factorial coagulopathy. Due to these circumstances, cardiac surgery patients account for up to 20% of total annual blood transfusion with a subset of high risk patients consuming 80% of all transfusion in this group. On this basis, employing blood conservation methods is extremely relevant as the use of donated blood products leads to greater rates of infectious complications, atrial fibrillation, prolonged postoperative ventilation, acute renal injury, and reduced short and long-term survival in cardiac surgery patients. Reducing the health and cost burden associated with transfusion is an important outcome to both the patient and health care system. Intraoperative autologous whole blood transfusion, a blood-conservation method similar to acute normovolemic hemodilution, may reduce transfusion and its associated complications but there is a paucity of large scale prospective randomized control trials investigating its efficacy in the era of modern surgical approaches, targeted transfusion using point-of-care viscoelastic testing, and advanced perfusion techniques. The intent of this study is to assess the feasibility of a trial protocol for a large-scale national study investigating high volume autologous whole blood transfusion for reduction in allogenic transfusion, derivative administration, and transfusion-associated morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 yr)
* Surgical patients at the Mazankowski Alberta Heart Institute
* High risk for acquired coagulopathy

Exclusion Criteria:

* Left ventricular ejection fraction <20%
* Impaired renal function
* Preoperative anemia (hematocrit < 30%)
* Abnormal coagulation studies or platelet function
* Presence of hemoglobinopathy
* Platelet count < 120 10*9/L
* Non-heparin based CPB anticoagulation
* Presence of carotid stenosis (≥70%)
* Presence of bacteremia/endocarditis
* Age > 85 yr
* Weight < 55 kg
* Hepatic failure/dysfunction
* Pregnancy
* Chronic lung disease on home O2
* Acute respiratory failure
* Acute coronary syndromes
* Emergency surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Adequacy of recruitment. | 12 months.
  Proportion of screened eligible patients that are successfully recruited.

SECONDARY OUTCOMES:
Number of allogenic units transfused. | 24 hours
  Number of units of red blood cell, plasma, platelets, cryoprecipitate administered intra-operatively and within the first 24hrs post-operatively.
Dose of prothrombin complex concentrates. | 24hrs
  Dose (in units per kilogram) of prothrombin complex concentrates given intraoperatively and within the first 24 hrs postoperatively.
Dose of fibrinogen. | 24 hrs
  Dose (grams per kilogram) of fibrinogen given intraoperatively and within the first 24 hrs postoperatively.
24-Hour chest tube output. | 24 hours
  Measured in millilitres during first 24 hours post-operatively.
Time to extubation. | 30 days
  Measured in hours from time of arrival to ICU admission (index admission) until extubated.
ICU length of stay. | 30 days
  Measured as number of days in ICU.
Hospital length of stay. | 30 days
  Measured as number of days in hospital.
Incidence of postoperative myocardial infarction (MI). | 30 days
  As measured by laboratory serum troponin and one or more of: new left bundle branch block, new pathological Q waves on electrocardiogram, new regional wall motion abnormality on echocardiogram, identification of intracoronary thrombus on angiography or at the time of autopsy.
Incidence of infection. | 30 days
  Any new infection following cardiac surgery and within the first 30 days post-operatively.
Incidence of post-operative stroke. | 30 days
  Defined as any acute onset focal neurological deficit lasting more than 24 hours that corresponded to clinical assessment and brain imaging.
Incidence of acute lung injury. | 30 days
  Defined as any acute inflammation in the lung that causes disruption of the lung endothelial and epithelial barriers with partial pressure of oxygen tension in arterial blood (PaO2) to fraction inspired oxygen (FiO2) ratio of less than 300.
Incidence of acute kidney injury (AKI). | 30 days
  Defined per the Kidney Disease Improving Global Outcomes (KDIGO ) criteria for Stage 2 and 3 AKI: 2.0-2.9 time postoperative increase in serum creatinine from preoperative value (stage 2); greater than 3.0 times increase in serum creatinine from preoperative value or increase in serum creatinine to greater than or equal to 353.6 micromole per litre or initiation of new renal replacement therapy postoperatively (stage 3) within 30 days.
Incidence of new requirement renal replacement therapy. | 30 days
  Defined as any new postoperative requirement of renal replacement therapy within the first 30 days of surgery.
Incidence of new onset atrial fibrillation. | 30 days
  Defined as new postoperative atrial fibrillation, persistent or paroxysmal, within the first 30 days postoperative.
Incidence of death within 30-days post-operatively. | 30 days
  Defined as death within the first 30 days postoperative.

OTHER OUTCOMES:
Research assistant cost per participant. | 12 months
  Assess time required of research assistant to enroll participant and extract data variables from electronic medical record.
Proportion of recruited participants successfully randomized. | 12 months
  Assess proportion of recruited participants that are successfully randomized with (target of >80%).
Number of participants with inadvertent unblinding of the intensive care clinicians. | 12 months
  Assess number of participants with inadvertent unblinding of the intensive care clinicians (target of <5%).
Number of major protocol deviations (adherence). | 12 months
  Assess number and define areas of protocol deviations.
Number of participants without complete follow-up. | 12 months
  Assess number of participants lost to follow-up (target <10%).

CONTACTS AND LOCATIONS:
Overall Officials: Angela R Neufeld, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada